CLINICAL TRIAL: NCT00999362
Title: Is T-lymphocyte Calcineurin Phosphatase Up-regulated by Treatment With Tacrolimus?
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Danish Society of Nephrology (Other); The Danish Kidney Association (Other); Astellas Pharma Inc (Industry)
Responsible Party: MD Dorthe M Mortensen, Department of Nephrology, Aarhus University Hospital, Skejby, Denmark
Other Study IDs: TAC
Record Dates: First submitted 2009-10-20; First posted 2009-10-21 (Estimated); Last update posted 2009-10-21 (Estimated); Status verified 2009-10

CONDITIONS: Kidney Transplantation
Keywords: calcineurin activity; real-time PCR; Gene expression of calcineurin; T-lymphocytes; interferon-gamma; Pharmacodynamics; Pharmacokinetics; tacrolimus; western blot; Hoechst

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Early kidney-transplant recipients: Patients receiving a kidney transplantation at Aarhus University Hospital, Skejby and receiving tacrolimus as part of their immunosuppressive regime.
- stable kidney transplant recipients: Tacrolimus treated kidney-transplant recipients from the out-door clinic at Aarhus University Hospital, Skejby and more than two years after transplantation

SUMMARY:
The purpose of this study is to determine whether calcineurin phosphatase in the T-lymphocytes is up-regulated after long-term treatment with tacrolimus, a calcineurin inhibitor.

DETAILED DESCRIPTION:
Background:

The immunosuppressive effect of both tacrolimus and cyclosporine is believed to be through inhibition of the enzyme calcineurin phosphatase (CaN) in T-lymphocytes. We have demonstrated, that tacrolimus decreases CaN activity in patients early after renal transplantation. In stable renal transplant patients treated this inhibition was hardly seen in patients treated with tacrolimus, while it was clearly demonstrated in patients treated cyclosporine. One explanation to this finding could be, that calcineurin phosphatase is up-regulated by long-term treatment with tacrolimus. The findings seem to imply, that tacrolimus has mechanisms of immunosuppression apart from inhibiting CaN. This could have implications for side-effects due to CaN inhibition. Among side-effects thought to be due to CaN inhibition is nephrotoxicity. The results may therefore be and indication of tacrolimus being less nephrotoxic compared to cyclosporine in long-term stable renal transplant patients.

Purpose:

The aim of the project is find out if long-term treatment with tacrolimus results in up-regulation of CaN in lymphocytes.

Study plan:

The general plan of the investigation is to compare CaN in lymphocytes in two groups of renal transplant patients treated with tacrolimus. One group just prior and just after transplantation compared to a group of stable renal transplanted patients a long time after transplantation. CaN is determined as enzyme activity, amount of protein, and by gen-activation.

ELIGIBILITY:
Inclusion Criteria:

Group 1 (early kidney-transplant recipients)

* Age over 18 years
* 20 consecutively kidney-transplant recipients at Department of Nephrology, Aarhus University Hospital, Skejby, Denmark
* receiving tacrolimus as part of their immunosuppressive treatment
* receipt of graft from either deceased or living-related donor
* written consent to participate

Group 2 (stable kidney-transplant recipients)

* Age over 18 years
* Stable renal allograft function defined as S-creatinine <200 µmol/l
* variation in S-creatinine <20% for 6 months prior to inclusion
* kidney transplantation more than 2 years before inclusion
* receipt of graft from either deceased or living-related donor
* written consent to participate

Exclusion Criteria:

Group 1 (early kidney-transplant recipients)

* patients suspected of non-compliance
* patients receiving medications known to interact with tacrolimus pharmacokinetics
* patients who on day 8 after transplantation have not reached a trough level for blood tacrolimus concentration above 8 µg/l.

Group 2 (stable kidney-transplant recipients)

* patients suspected of non-compliance
* patients receiving medications known to interact with tacrolimus pharmacokinetics

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Kidney transplant recipients from Department of Nephrology, Aarhus University Hospital, Skejby, Denmark
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2007-10; Primary Completion 2009-03 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Gene expression of calcineurin in T-lymphocytes | Trough level and 2 hours postdose
Calcineurin activity measured in whole blood and in isolated T-lymphocytes | Trough level and 2 hours postdose
Amount of Calcineurin in T-lymphocytes | Trough level and 2 hours postdose
Interferon-gamma production | Trough level and 2 hours postdose

SECONDARY OUTCOMES:
Tacrolimus concentration in whole blood | Trough level and 2 hours postdose
Number of T-lymphocytes | Trough level and 2 hours postdose

CONTACTS AND LOCATIONS:
Overall Officials: Dorthe M Mortensen, MD, Principal Investigator — Department of nephrology, Aarhus University Hospital,Skejby, Denmark
Locations (1):
- Department of Nephrology, Aarhus University Hospital, Skejby, Aarhus, Denmark